CLINICAL TRIAL: NCT06111157
Title: Clinical Spectrum of Infants of Diabetic Mothers , in Neonatal Intensive Care Unit of Assiut University Children's Hospital
Brief Title: Infants of Diabetic Mothers in Neonatology Unit at Assiut University Children's Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Nasser Mahrous Danial, Principle investigator, Assiut University
Other Study IDs: Infants of diabetic mothers
Record Dates: First submitted 2023-10-14; First posted 2023-11-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Infant of Diabetic Mother

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determine spectrum of clinical presentations and complications associated with maternal diabetes mellitus in their newborns attending and admitted to Neonatal Intensive Care Unit of Assiut University Children's Hospital.

DETAILED DESCRIPTION:
The global incidence of diabetes mellitus including diabetes of pregnant women is on the rise .

Diabetes during pregnancy has been associated with several maternal and fetal problems .

Diabetes during pregnancy include gestational diabetes which is defined as carbohydrate intolerance of varying degrees with hyperglycemia starting during pregnancy ,generally develops in the second half of pregnancy .

While pregestational diabetes is the condition in which a woman with diabetes ( type 1 or commonly type 2 ) before the onset of pregnancy .

Both gestational and pregestational diabetes are associated with increased rates of adverse maternal and neonatal outcomes . Adverse outcomes are more common with pregestational diabetes compared to gestational diabetes mellitus ; although , conflicting results have been reported .

Inspite the huge progress in the treatment of diabetes mellitus , Investigators are still in the situation that both gestational and pregestational diabetes impose an additional risk to the embryo , fetus , and course of pregnancy Pregestational diabetes mellitus increases the rate of congenital malformations , especially cardiac such as Patent foramen ovale , hypertrophic cardiomyopathy , Atrial septal defect , ventricular septal defect .

Fetal macrosomia is a common adverse effect on the infant outcomes . It increases the risk of shoulder dystocia , clavicle fractures , brachial plexus injury , which increase the rate of admission to the neonatal intensive care unit .

This infant may experience asphyxia , respiratory distress , hypoglycemia or hyperglycemia , hyperinsulinemia , hypocalcemia , hypomagnesemia , hyperbilirubinemia , polycythemia and anemia .

Caudal regression syndrome , anencephaly , microcephaly , hydrocephalus , spina bifida are also complications of diabetes mellitus in pregnancy .

Both gestational and pregestational diabetes may also cause various motor and behaviouralneurodevelopmental problems including an increased incidence of attention deficit hyperactivity disorder and autism spectrum disorder .

It has been found that there is increased rate of obesity , impaired glucose intolerance or diabetes mellitus in the childhood and adolescence .

Mechanisms of diabetic induced damage in pregnancyare related to maternal and fetal hyperglycemia ,enhanced oxidation status , epigenetic changes and other less defined pathogenic mechanisms .

Uncontrolled diabetes has profound effects on embryogenesis , organogenesis , and fetal and neonatal growth .

The severity of complications is higher with earlier onset of gestational diabetes mellitus and inversely correlated with the degree of glycemic control .

Early initiation of gestational diabetes mellitus might even cause some increase in the rate of congenital malformations .

Tight glycemic control prior to conception and during pregnancy can prevent an excess rate of congenital malformations ,macrosomia , birth trauma and neonatal respiratory distress syndrome .

ELIGIBILITY:
Inclusion Criteria:

* The study will include all live births of diabetic mothers attending and admitted to Neonatal intensive Care Unit of Assiut University Children's Hospital .

Exclusion Criteria:

* Babies born to non diabetic mothers .

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include all live births of diabetic mothers attending and admitted to Neonatal intensive Care Unit of Assiut University Children's Hospital .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Determine clinical spectrum of infants of diabetic mothers at neonatology unit of Assiut university children's hospital | Baseline
  Mesure weight in kelograms
Determine clinical spectrum of infants of diabetic mothers | baseline
  Mesure height in centimeters
Determine clinical spectrum of infants of diabetic mothers | baseline
  Mesure head circumference in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Safwat Mohamed Abdel-aziz, Assistant professor, Study Director — Assiut University; Shimaa Kamal Mohamed, Lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Singh S, Yadav M. Gestational Diabetes Mellitus among Pregnant Women Delivering in a Tertiary Care Hospital: A Descriptive Cross-sectional Study. JNMA J Nepal Med Assoc. 2022 Mar 11;60(247):229-233. doi: 10.31729/jnma.7304. PMID 35633259
- [Background] Ornoy A, Becker M, Weinstein-Fudim L, Ergaz Z. Diabetes during Pregnancy: A Maternal Disease Complicating the Course of Pregnancy with Long-Term Deleterious Effects on the Offspring. A Clinical Review. Int J Mol Sci. 2021 Mar 15;22(6):2965. doi: 10.3390/ijms22062965. PMID 33803995
- [Background] Malaza N, Masete M, Adam S, Dias S, Nyawo T, Pheiffer C. A Systematic Review to Compare Adverse Pregnancy Outcomes in Women with Pregestational Diabetes and Gestational Diabetes. Int J Environ Res Public Health. 2022 Aug 31;19(17):10846. doi: 10.3390/ijerph191710846. PMID 36078559
- [Background] Akbariasbagh P, Shariat M, Akbariasbagh N, Ebrahim B. Cardiovascular Malformations in Infants of Diabetic Mothers: A Retrospective Case-Control Study. Acta Med Iran. 2017 Feb;55(2):103-108. PMID 28282706
- [Background] Kc K, Shakya S, Zhang H. Gestational diabetes mellitus and macrosomia: a literature review. Ann Nutr Metab. 2015;66 Suppl 2:14-20. doi: 10.1159/000371628. Epub 2015 Jun 2. PMID 26045324
- [Background] Weintrob N, Karp M, Hod M. Short- and long-range complications in offspring of diabetic mothers. J Diabetes Complications. 1996 Sep-Oct;10(5):294-301. doi: 10.1016/1056-8727(95)00080-1. PMID 8887019
- [Background] [7] J. L. Kitzmiller, A. Ferrara, T. Peng, M. A. Cissell, and C. Kim, "Chapter 5: Preexisting Diabetes and Pregnancy."